CLINICAL TRIAL: NCT02811016
Title: Effect of Inhaled Budesonide on the Incidence and Severity of Acute Mountain Sickness at 4559 m
Brief Title: Inhaled Budesonide and Acute Mountain Sickness
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Salzburger Landeskliniken (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Principal Investigator, Marc Berger, PD Dr. med., Salzburger Landeskliniken
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M2016
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Acute Mountain Sickness
Keywords: High Altitude; budesonide; hypoxia
MeSH Terms: conditions — Altitude Sickness; Hypoxia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- budesonide 200 (Experimental): inhaled budesonide 200 µg bid
  Interventions: Drug: Budesonide 200
- budesonide 800 (Experimental): inhaled budesonide 800 µg bid
  Interventions: Drug: Budesonide 800
- placebo (Placebo Comparator): inhaled placebo bid
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Budesonide 200 — 200 µg inhaled at 7:00 a.m. and 7 p.m.
  Other Names: Pulmicort Turbohaler
  Arms: budesonide 200
Drug: Budesonide 800 — 800 µg inhaled at 7:00 a.m. and 7 p.m.
  Other Names: Pulmicort Turbohaler
  Arms: budesonide 800
Drug: Placebo — Placebo Inhalation at 7:00 a.m. and 7 p.m.
  Other Names: Lactose-Monohydrate
  Arms: placebo

SUMMARY:
The primary objective of the study is to investigate the effect of inhaled budesonide on the incidence of AMS. The primary study question to ask is:

1. Does inhaled budesonide reduce the incidence of AMS after rapid and active ascent to 4559 m?

In addition, the secondary study questions to ask are:

1. Does inhaled budesonide reduce the severity of AMS after rapid and active ascent to 4559 m?
2. Are the effects of inhaled budesonide on AMS incidence and severity related to its plasma concentration?

Study medication Inhaled budesonide at 2 different concentrations (2 x 200 µg, 2 x 800 µg) versus placebo

Study design

* Prospective, controlled, single-center study on 51 healthy volunteers at 4559 m [Capanna Regina Margherita (Margherita Hut), Italy]
* With regard to the intervention (inhaled budesonide) double-blinded and randomized

DETAILED DESCRIPTION:
Primary objective

The primary objective of the study is to investigate the effect of inhaled budesonide on the incidence of AMS. The primary study question to ask is:

1. Does inhaled budesonide reduce the incidence of AMS after rapid and active ascent to 4559 m?

In addition, the secondary study questions to ask are:

1. Does inhaled budesonide reduce the severity of AMS after rapid and active ascent to 4559 m?
2. Are the effects of inhaled budesonide on AMS incidence and severity related to its plasma concentration?

Study medication Inhaled budesonide at 2 different concentrations (2 x 200 µg, 2 x 800 µg) versus placebo

Study design Prospective, controlled, single-center study on 51 healthy volunteers at 4559 m [Capanna Regina Margherita (Margherita Hut), Italy] With regard to the intervention (inhaled budensoide) double-blinded and randomized

Study population 51 healthy volunteers

Study site Prior to the study the pre-investigations will be performed at the University Hospital Salzburg, Austria. The high-altitude part will take place at the Capanna Regina Margherita (Margherita Hut, Italy) at 4559 m.

Interventions and investigations

* Ascend from Alagna (1130 m, Italy) to the Margherita Hut (4559 m) in less than 24 h, with a preceding overnight stay at 3611 m (Gnifetti Hut, Italy).
* Stay at the Margherita Hut for 48 hours
* Randomized inhalation of budesonide at two different concentrations (2 x 200 µg 2 x 800 µg, respectively) or placebo
* Assessment of incidence and severity of acute mountain sickness by use of 2 internationally standardized and well established questionnaires
* Venous (and capillary) blood drawings
* Pulmonary function tests
* Transthoracic echocardiography for assessing pulmonary artery systolic pressure

Number and volume of blood drawings For the study venous blood samples (volume: 20 ml each) will be drawn at 5 different time points (5 x 20 ml = 100 ml). Together with the blood drawing for the pre-investigation (20 ml) a total blood volume of 120 ml will be taken. At the same time points capillary blood samples (1 ml) will be taken from the ear lobe for blood gas analyses (5 x 1 ml = 5 ml in total).

Observational period The study will only start after approval by the ethic committee responsible for the study (ethic committee of the Paracelsus Medical University). If the study is approved it will be performed in July 2016.

ELIGIBILITY:
Inclusion Criteria:

* Good physical condition
* No relevant pathologies revealed by the pre-investigation prior to the study
* Written informed consent to participate in the study
* Permanent residency below 1000 m
* Males and females are included without prioritization

Exclusion Criteria:

* Acute and chronic lung diseases
* Conventional systolic blood pressure (average of two measurements) ≥150 mmHg and conventional diastolic blood pressure ≥95 mmHg in untreated or treated subjects
* Cardiovascular diseases other than hypertension (coronary heart disease, heart failure, atrial fibrillation, peripheral artery disease)
* Chronic headache / migraine
* Diabetes mellitus
* Smoking (>6 cigarettes/day) or equivalent nicotine substitutes
* Alcohol (>30 g/d) or drug abuse
* Obesity (Body Mass Index >30)
* Other conditions deemed relevant by the investigator (including liver disease, renal disease)
* Sojourn >2000 m within the last 4 weeks before the 1st study day
* Drug intake within the last 2 moth before the 1st study day if the drug intake could affect the data quality or the safety of the participants
* Blood donation within the last 2 month before the 1st study day

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2016-06; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Incidence of acute mountain sickness | 48 hrs at 4559 m
  AMS scores positive

SECONDARY OUTCOMES:
Severity of acute mountain sickness | 48 hrs at 4559 m
  Height of AMS scores

CONTACTS AND LOCATIONS:
Overall Officials: Marc M Berger, MD, Principal Investigator — Department of Anesthesiology, University Hospital Salzburg
Locations (1):
- Department of Anesthesiology, University Hospital, Salzburg, Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger MM, Macholz F, Sareban M, Schmidt P, Fried S, Dankl D, Niebauer J, Bartsch P, Mairbaurl H. Inhaled budesonide does not prevent acute mountain sickness after rapid ascent to 4559 m. Eur Respir J. 2017 Sep 10;50(3):1700982. doi: 10.1183/13993003.00982-2017. Print 2017 Sep. No abstract available. PMID 28890439